CLINICAL TRIAL: NCT04697602
Title: Low-dose Colchicine With or Without Stepwise Dose Titration of Febuxostat for Flare Prophylaxis in Patients With Gout and Hyperuricemia During the Initial Phase of Urate-lowering Therapy: an Open-label Randomized Controlled Trial
Brief Title: Low-dose Colchicine With or Without Stepwise Dose Titration of Febuxostat for Flare Prophylaxis in Gout
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202009131MIND
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Gout
Keywords: gout,febuxostat,flare prophylaxis,stepwise dose titration,colchicine
MeSH Terms: conditions — Gout | interventions — Colchicine; Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose titration group (Experimental): Stepwise dose titration of febuxostat and low-dose colchicine
  Interventions: Drug: Stepwise dose titration of febuxostat and low-dose colchicine
- Standard treatment group (Active Comparator): Fixed dose febuxostat and low-dose colchicine
  Interventions: Drug: Fixed dose febuxostat and low-dose colchicine

INTERVENTIONS:
Drug: Stepwise dose titration of febuxostat and low-dose colchicine — Febuxostat 10 mg, orally, once daily, in week 1-4 Febuxostat 20 mg, orally, once daily, in week 5-8 Febuxostat 40 mg, orally, once daily, in week 9-12 Concomitant colchicine 0.5 mg, orally, once daily in week 1-12
  Arms: Dose titration group
Drug: Fixed dose febuxostat and low-dose colchicine — Febuxostat 40 mg, orally, once daily, in week 1-12 Concomitant colchicine 0.5 mg, orally, once daily in week 1-12
  Arms: Standard treatment group

SUMMARY:
The purpose of this study is to compare the incidence rate of gout flare for subjects with gout and hyperuricemia treated by two different starting doses of febuxostat.

DETAILED DESCRIPTION:
A prospective randomized open-label study comparing dose titration group (stepwise dose titration of febuxostat and low-dose colchicine) and standard treatment group (fixed dose febuxostat and low-dose colchicine) in the subjects with gout and hyperuricemia. The incidence rate of gout flare will be compared between two groups during the first 12 week of febuxostat treatment.

ELIGIBILITY:
Ages Eligible for Study: more than 20 years

Inclusion Criteria:

1. Hyperuricemia (serum urate ≥7.0 mg/dL and gout by 1977 American College of Rheumatology Criteria
2. Acute gout attack during the last 12 months

Exclusion Criteria:

1. Acute gout attack in the last 2 weeks
2. Urate-lowering therapy in the last 4 weeks
3. Secondary hyperuricemia
4. Creatinine ≥2.0 mg/dL
5. AST or ALT ≥2x upper limits of normal
6. Heart failure (NYHA III-IV)
7. Hypersensitivity to colchicine, NSAID or febuxostat
8. Use of NSAID, glucocorticoid, cyclosporine, clarithromycin, mercaptopurine, azathioprine, pyrazinamide, ethambutol, chemotherapy, tacrolimus, losartan, and fenofibrate
9. Inability to comply with the protocol requirements
10. The judgement of the investigator that the patient was not an appropriate candidate

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
The incidence rate of gout flare during the first 12 weeks. | 12 weeks
  The percentage of the patients suffered from gout flare during the first 12 weeks.

SECONDARY OUTCOMES:
The number of gout flares per patient during the first 12 weeks | 12 weeks
  The number of gout flares per patient during the first 12 weeks
The number of gout flares per patient during the second 12 weeks | 12 weeks
  The number of gout flares per patient during the second 12 weeks
The percentage of patients with serum urate <6.0mg/dL in 12, 24 weeks | 12, 24 weeks
  The percentage of patients with serum urate <6.0mg/dL in 12, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Min Huang, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan